CLINICAL TRIAL: NCT03989687
Title: Clinical Retention of Glass Ionomer Sealants Placed With and Without Rubber Dam: a Comparative Analysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Suzanne E Fournier, Assistant Professor, Louisiana State University Health Sciences Center in New Orleans
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 19-138
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Dental Caries in Children

STUDY DESIGN:
Intervention Model Description: each patient is serving as their own control
Who Masked: Outcomes Assessor
Masking Description: The evaluator will not have knowledge of which type of isolation was used when placing the sealants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- glass ionomer sealant (Experimental): glass ionomer sealant
  Interventions: Other: isolation
- isolation (Experimental): isolation type either rubber dam or cotton roll isolation
  Interventions: Device: Fuji Triage

INTERVENTIONS:
Device: Fuji Triage — glass ionomer sealant
  Other Names: Fuji VII
  Arms: isolation
Other: isolation — rubber dam or cotton roll isolation
  Arms: glass ionomer sealant

SUMMARY:
A comparative analysis of glass ionomer sealant placed on permanent molars with and without a rubber dam to assess the retention over a 2 year period.

DETAILED DESCRIPTION:
The purpose of the study is to compare the retention rates of glass ionomer sealants placed on first permanent molars over a period of 2 years. Pediatric patients (under <10 years of age) will receive a glass ionomer sealant on all four permanent first molars. One side will be randomly selected with rubber dam isolation and the contralateral side will have no rubber dam isolation for the placement of the sealant. Over a 2 year period, every 6 months the sealants will be assessed for retention.

The glass ionomer sealant material will be Fuji Triage (GC America). The following dental materials that will be used are cotton rolls, non-latex rubber dam, topical benzocaine, dental mirror, glass ionomer dispensing gun, dental explorer, triturator for the glass ionomer, cotton gauze, suction tip, air-water syringe.

ELIGIBILITY:
Inclusion Criteria: healthy children who need sealants on 4 permanent molars that are not hypo plastic, are caries-free, and with no enamel defects.

-

Exclusion Criteria: hypoplastic molars, caries, teeth with existing restorations, and those with enamel defects,

-

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
retention rate of sealants | 6 months
  retention rate for sealants placed with different modes of isolation

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Fournier, DDS, Principal Investigator — LSUHSC

IPD SHARING:
Plan to Share IPD: No